CLINICAL TRIAL: NCT00657072
Title: Biomechanical Evaluation of Wrist Ligament Injuries: Diagnostic Tool to Detect Wrist Instability
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Walter H. Short, M.D., SUNY Upstate Medical University
Other Study IDs: 4840; 1R01AR050099 (NIH)
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-11

CONDITIONS: Scapholunate Interosseous Ligament; Torn Wrist Ligaments
Keywords: scapholunate instability; neural networks; scaphoid; lunate; Suspected torn scapholunate interosseous ligament; Suspected other torn wrist ligaments

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Damage to the ligaments of the wrist occurs frequently, however, it is not well publicized or understood. Our previous and current biomechanical studies have shown that damage to certain wrist ligaments is the likely cause of wrist instability and pain. Based on our three dimensional models and animations of actual cadaver motions with various ligaments intact or sectioned, we have identified several changes in how the carpal bones move and are positioned relative to the radius with various levels of instability. Using this information, we have developed a mathematical model that can predict in cadaver wrists which groups of ligaments have been injured. We started, under IRB approval, a prospective clinical study to evaluate the reliability of this mathematical model. During the past 5 years we have studied 13 patients with suspected wrist ligament injuries who were previously scheduled for surgical treatment. CT scans have been performed of the injured wrist and for comparison purposes, the contralateral, uninjured wrist. During these 5 years, there were no problems with the conduct of the study. During these 5 years the only changes to the original study application were

* a) to include a CT scan of the contralateral wrist for comparison purposes
* b) a paper handout given to potential subjects
* c) to add additional people to the study team.

The principal investigator, blinded to the results of the CT scan, surgically explores and treats these patients in the same manner that he would for any patient with suspected wrist ligament injuries. During the surgery, the investigator determines the integrity of the various wrist ligaments. The prediction of which ligaments are damaged, based upon the CT scan information and mathematical model is compared to the actual surgical findings. The importance of this study is to develop a tool that will allow one to rapidly and non invasively diagnose wrist instability and initiate treatment before further damage is done.

ELIGIBILITY:
Inclusion Criteria:

* patients who have suffered ligamentous injuries to their wrists and have been referred to the principal investigator
* subject selected to undergo surgery
* The ethnicity and racial makeup of the group is similar to the demographics of the surrounding referral base
* There will be no exclusion of any gender, racial or ethnic group

Exclusion Criteria:

* Pregnant women will not be included because of increased anesthetic risks at surgery.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients who have suffered ligamentous injuries to their wrists will be recruited for this study
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2003-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter H Short, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Musculoskeletal Science Research Center, Syracuse, New York, United States